CLINICAL TRIAL: NCT07049497
Title: Monocentric Retrospective Observational Study on Immune Response in Biological Samples Belonging to Subjects Vaccinated Against SARS-CoV-2 Infection
Brief Title: Study of Immune Response in Subjects Vaccinated Against SARS-CoV-2 Infection
Acronym: BioVAC-immunit
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Rovere Querini Patrizia, MD, PhD, IRCCS San Raffaele
Other Study IDs: BioVAC-immunity
Record Dates: First submitted 2025-06-25; First posted 2025-07-03 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-06

CONDITIONS: SAR-CoV-2; Cellular Immune Response; Antibody Response

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Aliquots of PBMC collected at the completion of the vaccination cycle and frozen at the CRB
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 107 healthcare workers who completed the vaccination cycle for SARS-CoV-2: T cell response in terms of IFN-γ measured by ELISpot
  Interventions: Other: Evaluation of the T cell response in terms of IFN-γ measured by ELISpot
- 20 healthy donors who didn't receive SARS-CoV-2 vaccination: T cell response in terms of IFN-γ measured by ELISpot
  Interventions: Other: Evaluation of the T cell response in terms of IFN-γ measured by ELISpot

INTERVENTIONS:
Other: Evaluation of the T cell response in terms of IFN-γ measured by ELISpot — The evaluation of the T cell response will be performed by quantifying the frequencies of SARS-CoV-2-specific T cells producing IFN-γ using an enzyme-linked immunospot assay (ELISpot), with cryopreserved PBMC collected at the designated timepoints (T0, T1, T2, T3, and T4)

SUMMARY:
Twelve months after the first SARS-CoV-2 cases in Wuhan, the FDA approved the first COVID-19 vaccine (Pfizer-BioNTech). Early studies on healthcare workers showed that antibody levels, especially against the Spike protein, declined within six months, particularly in those without prior infection. However, previously infected individuals had stronger and longer-lasting responses. The vaccine induces a Th1-type T cell response, linked to milder disease, and activates follicular helper T cells and B cell responses, although antibody levels drop over time. Immune responses also differ by sex, with females showing stronger humoral responses. Key priorities include understanding humoral fluctuations, characterizing cellular immunity, and correlating both responses.

ELIGIBILITY:
healthcare workers group

Inclusion Criteria:

* Male and/or female sex

Age ≥18 years

Completion of the SARS-CoV-2 vaccination cycle with the Pfizer-BioNTech vaccine

Informed consent for the storage of biological material at the San Raffaele Hospital Biological Resource Center (with protocol related to the BioVAC study approved by the Ethics Committee: 17/INT/2022)

Availability of at least two aliquots of PBMC collected at the completion of the vaccination cycle and frozen at the CRB

Exclusion Criteria:

* none donor group

Inclusion Criteria:

- consent for sample collection and storage in the Biobank between 2016 and 2018

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Approximately 405 biological samples will be analyzed in the study, collected from the OSR Biobank (with protocol related to the BioVAC study approved by the Ethics Committee: 17/INT/2022). These samples were obtained from healthcare workers who completed the SARS-CoV-2 vaccination cycle between January 2020 and November 2021.
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2022-06-28 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
To assess the existence of a correlation between the antibody titer six months after the second dose and the T and B cell responses | Six months after the second vaccine dose, which coincides with the time of enrollment
  Correlation between antibody titer, in terms of antibodies directed against the Spike protein, and T cell response, in terms of IFN-γ measured by ELISpot, as well as B cell response, in terms of frequency and phenotype, assessed six months after the second dose (T3)

CONTACTS AND LOCATIONS:
Overall Officials: Patrizia Rovere Querini, PhD, MD, Principal Investigator — IRCCS Ospedale San Raffaele
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Italy, Italy

IPD SHARING:
Plan to Share IPD: No